CLINICAL TRIAL: NCT06575348
Title: Implementation of the YouControl-AFib mHealth Application (Pilot Version) to Improve Physical Activity in Persons With Atrial Fibrillation
Brief Title: Evaluation of YouControl-AFib, a mHealth Application for Persons With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0954; A534225 (Other: UW Madison); Protocol Version 8/6/2024 (Other: UW Madison); 1UL1TR002373 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: physical exercise; application; supportive care
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- People using YouControl-A-Fib app (Experimental)
  Interventions: Device: YouControl-A-Fib mHealth Application

INTERVENTIONS:
Device: YouControl-A-Fib mHealth Application — Participants will use the app for 3 months, includes 1 month phone call with Health Coach

SUMMARY:
This study is being done to establish the feasibility of performing a clinical trial using a mHealth application named YouControl-AFib designed to improve the cardiovascular health of persons with atrial fibrillation. The study will obtain feedback on the app design to inform future versions and will collect preliminary data to support proof-of-concept and potential effect sizes for future trial design.

DETAILED DESCRIPTION:
Primary Objective

* To effectively recruit participants for a clinical trial and obtain user feedback on the mHealth app using the Mobile App Rating Scale and focus group sessions.

Secondary Objectives

* To evaluate the impact of the YouControl-AFib mHealth app (pilot version, 3 months of use) on physical activity in persons with atrial fibrillation.
* To obtain several additional functional and disease specific endpoints that will help establish possible effect sizes to be evaluated more formally in subsequent versions of the mHealth application.
* To obtain user feedback on the mHealth app using the Mobile App Rating Scale and focus group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Willing to comply with all study procedures and be available for the duration of the study
* SmartPhone capable of pairing with a Fitbit Sense 2 and Fitbit App (Apple iOS 15 and higher or Android 10 or higher)
* Paroxysmal or persistent atrial fibrillation verified by 12-lead electrocardiogram (ECG) or other clinical grade monitoring
* body mass index (BMI) greater than 27

Exclusion Criteria:

* History of permanent atrial fibrillation
* Left ventricular ejection fraction (LVEF) less than 45 percent
* Myocardial infarction, coronary artery bypass grafting, or valve surgery within the last 12 months
* Moderate to severe valve disease
* Inability to participate in a structured exercise program due to musculoskeletal disease
* Already participating in a structured exercise program or achieving guideline directed physical activity
* Planned surgery or procedure during the next three months that limit ability to engage in physical activity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Average Number of Participants Recruited Per Month | up to 5 months
Maximum Number of Participants Recruited Per Month | up to 5 months
Mobile App Rating Scale Scores | 3 months
  Mobile App Rating Scale contains several subscales that will each be scored on a scale of 1-5; B-functionality, C-aesthetics, and D-information. Higher scores indicate high levels of functionality, aesthetics, and information quality.

SECONDARY OUTCOMES:
Change in 6-minute walk distance (compared to baseline for each participant) after using the mHealth app for 3 months | baseline, 3 months
Change in daily step count (averaged over 7 days) after using the mHealth app for three months | baseline, 3 months
Change in intentional activity time (in one week) after using the mHealth app for three months | baseline, 3 months
Change in general quality of life questionnaire: SF-12 Score | baseline, 3 months
  SF-12 measures the impact of health on the participant's life and is scored from 0-100 where higher scores indicates higher health related quality of life.
Change in Patient Health Questionnaire (PHQ-9) Score | baseline, 3 months
  PHQ-9 is a 9-item questionnaire scored on a 4 point likert scale from 0-3 for a total possible range of scores from 0-27. Higher scores indicate increased depression.
Change in Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT) Score | baseline, 3 months
  AFEQT is a 20-item survey scored on a 7 point likert scale from 1-7 where higher scores indicate higher effect that atrial fibrillation has on the participant's quality of life.
Change in Atrial Fibrillation Symptom Severity (AFSS) Score | baseline, 3 months
  AFSS is a 7-item survey scored on a likert scale from 0-5 for a total possible range of scores from 0-35 where higher scores indicate greater symptom severity.
Change in Atrial Fibrillation Knowledge Assessment Tool (AFKAT) Score | baseline, 3 months
  AFKAT is a 21-item true / false assessment that measures knowledge about atrial fibrillation. Correct answers are scored with a 1 for a total possible range of scores from 0-21. Higher scores indicate increased knowledge of atrial fibrillation.
Change in the Life's Essential 8 score after using the mHealth app for three months | baseline, 3 months
  Life's Essential 8 score (LE8) is a composite score between 0-100 that assesses a participant's adherence to 8 lifestyle recommendations with improve cardiovascular health: diet, physical activity, smoking habits, body mass index, cholesterol, blood glucose, and sleep duration. Higher scores are indicative of higher adherence to healthy lifestyle.
Change in irregular heart rate notifications (in one week) after using the mHealth app for three months | baseline, 3 months
Change in ECG-age after using the mHealth app for three months | baseline, 3 months
  Participants will obtain single-lead ECGs at baseline and after three months. The time-voltage data are run through an ECG-AI model for estimating ECG-age. ECG-age is a novel metric developed by investigators at Wake Forest. See reference section for relevant publication describing a similar model. Summary results will be reported as ECG-age in years.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Kalscheur, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. Every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers 7 years after the completion of the primary endpoint by contacting the PI.

REFERENCES:
- [Background] Attia ZI, Friedman PA, Noseworthy PA, Lopez-Jimenez F, Ladewig DJ, Satam G, Pellikka PA, Munger TM, Asirvatham SJ, Scott CG, Carter RE, Kapa S. Age and Sex Estimation Using Artificial Intelligence From Standard 12-Lead ECGs. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007284. doi: 10.1161/CIRCEP.119.007284. Epub 2019 Aug 27. PMID 31450977